CLINICAL TRIAL: NCT03401554
Title: Titanium Mesh Versus Collagen Membrane for Closure of Lateral Window Approach in Maxillary Sinus Floor Elevation With Simultaneous Implant Placement. Randomized Controlled Clinical Trial
Brief Title: Titanium Mesh Versus Collagen Membrane for Closure of Window in Maxillary Sinus Elevation With Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa mahmoud abd el fattah, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC.CU6.1.2018
Record Dates: First submitted 2018-01-06; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collagen membrane group (Active Comparator): Sinus floor elevation with simultaneous implant placement and closure of the osteotomy with collagen membrane
  Interventions: Procedure: collagen membrane
- titanium mesh group (Experimental): Sinus floor elevation with simultaneous implant placement and closure of the osteotomy with titanium mesh
  Interventions: Procedure: titanium mesh

INTERVENTIONS:
Procedure: titanium mesh — closing the lateral window for maxillary sinus floor elevation with titanium mesh
  Arms: titanium mesh group
Procedure: collagen membrane — closing the lateral window for maxillary sinus floor elevaion with collagen membrane
  Arms: collagen membrane group

SUMMARY:
Evaluation the amount of bone height gained when using titanium mesh in closing the lateral window of the sinus compared to collagen membrane.Evaluation the quality of new bone gained when using of the titanium mesh to close the lateral window of the maxillary sinus as a new option for tenting compared to collagen membrane.

DETAILED DESCRIPTION:
this study is aimed to review the bone height, quality and closure of lateral osteotomy used for maxillary sinus floor lifting comparing titanium mesh to collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* no signs of sinus pathology non or light smokers less than 20 cigarettes per day no systemic disease that may affect normal healing no pscychiatric problems no history of neoplasms or radiation therapy to the head and neck no previous bone augmentation to implant site

Exclusion Criteria:

* Sinus pathology. Heavy smokers more than 20 cigarettes per day Patients with systemic disease that may affect normal healing. Psychiatric problems Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-13 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
bone height | 6 months
  Evaluation the amount of bone height gained when using titanium mesh in closing the lateral window of the sinus compared to collagen membrane .

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mahmoud, Bds, Principal Investigator — Study principal investigator
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, الجيزة, Egypt